CLINICAL TRIAL: NCT04868097
Title: Predicting the Presence of Histologic Criteria for Adjuvant Post-operative Radiation of Patients With Cervical Cancer Stage IB2 by Large Loop Biopsy Prior to Surgery
Brief Title: Predicting Adjuvant Post-operative Radiation Therapy in Patients With Cervical Cancer Stage IB2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Collaborators: Barzilai Medical Center (Other); Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Alon Ben Arie, Director of obstetrics and gynecology department, Kaplan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0186-20-KMC; 0186-20-KMC (Other: Kaplan Medical Center)
Record Dates: First submitted 2021-04-26; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Cancer of the Cervix; Conization of the Cervix; Radiation Therapy
Keywords: cervix cancer, Radiation
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cervix biopsy — large loop electrosurgical cervix biopsy

SUMMARY:
A pre- operative evaluation for the presence of intermediate risk factors prior to surgery may allow for better patient counselling, modify the course of surgery or select patients to undergo primary chemo- radiation.

The purpose of this study is to validate that the presence of histological risk factors in a pre-operative large loop biopsy highly correlates with post-operative histological evaluation and the subsequent indication for post-operative chemo-radiation

DETAILED DESCRIPTION:
Patients with cervical cancer who are scheduled for radical hysterectomy and underwent a pre- operative MRI and PET- CT that have demonstrated a tumor ≥2- 4cm cm and the absence of nodal metastasis on imaging will be offered to give consent and participate.

After anesthesia and immediately prior to surgery, the surgeon will perform a large loop biopsy of depth of 1.5 and a diameter of 1.0 cm from the cervical tumor. Hemostasis can be achieved by the usual measures or by packing. Surgery will follow immediately as planned.

In patient who in the course of the preoperative evaluation underwent large loop biopsy histologic analysis of this biopsy will be performed similarly. If the large loop specimen is appropriate (>1.5X1cm) and allows assessment of all the histologic risk factors, no repeat large loop biopsy will be performed.

In patient that the that the previous large loop biopsy is not be appropriate for complete histologic analysis and the surgeon asses that a repeat biopsy is technically feasible, a large loop biopsy will be performed prior to the radical hysterectomy as described above.

All histological evaluation will be carried out as usual in hospital in which the surgery was performed.

In addition, centralized pathological analysis will be performed in Hillel Yaffe Medical center The histopathological features to be included in the report: type of procedure, tumor site, histologic type of tumor, histologic grade, depth of stromal invasion, pattern of invasion (*), horizontal extent of stromal invasion, the distance of tumor from surgical margins, lymphovascular invasion, LVSI will be assess and reported after D2-40and CD31 immunostatins.

Descriptive demographic, clinical and pathology data will be noted. The histopathological features noted above and size of tumor as measured on MRI will be recorded.

The rate of the presence of both LVSI and invasion greater 10 mm in the pre- operative loop biopsy will be assessed.

At least 52 patients will be included in the study

Sample size calculation:

The minimal sample size required to demonstrate the non-inferiority of Method B (findings in LEEP) is 52. Assuming that the proportions of patients with the presence of both LVSI and tumor invasion greater than 10 mm, method A (standard post- surgery evaluation) and method B are 25%, with α=0.05, β=0.2, and non-inferiority margin of 15%.

ELIGIBILITY:
1. Patients with cervical cancer who are scheduled for radical hysterectomy and underwent a pre- operative imaging (MRI and PET CT) that have demonstrated a tumor ≥2-4 cm and the absence of nodal metastasis.
2. Pre -operative assessment by the surgeon that a large loop biopsy of depth of 1.5 and a diameter of 1 cm is technically feasible.
3. Patient who in the course of the preoperative evaluation underwent large loop biopsy of depth of 1.5 and a diameter of 1.0 cm, and in the subsequent evaluation fulfilled the criteria in (1).

Exclusion Criteria:

Patient who do not sign the informed consent. Patient who is scheduled for Chemoradiation Patients with large loop biopsy which is smaller than depth of 1.5 and a diameter of 1.0 cm

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
The rate of LVSI in Cervix cancer | two years
  Pre operative presence of LVSI in loop biopsy in cervical cancer, compared to post operative LVSI rate in hysterectomy Specimen

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: No